CLINICAL TRIAL: NCT05347524
Title: Detection of Peritoneal Metastasis of Gastric Cancer by Liquid Biopsy in Peripheral Blood: A Prospective Study
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Guangzhou Burning Rock Bioengineering Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: B2022-081R
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Cancer
Keywords: stomach neoplasms; peritoneal metastasis; liquid biopsy; cell-free DNA (cfDNA) methylation
MeSH Terms: conditions — Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case arm - Gastric cancer with peritoneal metastasis: Baseline blood samples will be collected from gastric cancer participants with peritoneal metastasis.
  Interventions: Other: Baseline blood draw and blood-based biomarkers analyses
- Control arm - Gastric cancer without peritoneal metastasis: Baseline blood samples will be collected from gastric cancer participants without peritoneal metastasis.
  Interventions: Other: Baseline blood draw and blood-based biomarkers analyses

INTERVENTIONS:
Other: Baseline blood draw and blood-based biomarkers analyses — Baseline blood draw and blood-based biomarkers analyses

SUMMARY:
This study is a prospective, multi-omics, observational study aimed at detecting peritoneal metastasis of gastric cancer by combined assays for methylation of cell-free DNA (cfDNA) and other blood-based biomarkers. The study will enroll 384 participants with gastric cancer.

DETAILED DESCRIPTION:
Peritoneal metastasis (PM) in gastric cancer is associated with a poor prognosis.

Laparoscopy with cytology is performed to evaluate for peritoneal spread when considering chemoradiation or surgery. However, the laparoscopy is invasive and the sensitivity of computed tomography (CT) scan is poor for detecting PM. Therefore, it is necessary to evaluate the feasibility of cfDNA methylation and other blood-based biomarkers for the PM diagnosis.

The study will enroll 384 participants with gastric cancer. Baseline blood and diagnosis of PM by laparoscopy with cytology will be collected. Participants with PM will be defined as the case arm and participants without PM will be defined as the control arm. A PM diagnostic model will be developed.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for Case Arm Participants:

  1. Age 18-74 years at the day of consenting to the study.
  2. Able to provide a written informed consent.
  3. No prior cancer treatment (local or systematic) with either of the following:

     A. Pathologically confirmed gastric cancer diagnosis within 42 days prior to blood draw.

     B. High suspicious for cancer diagnosis by imaging tests or other routine clinical examinations, with confirmed pathological cancer diagnosis within 42 days after the blood draw.
  4. Diagnosis of peritoneal metastasis by laparoscopy with cytology.
* Inclusion Criteria for Control Arm Participants:

  1. Age 18-74 years at the day of consenting to the study.
  2. Able to provide a written informed consent.
  3. No prior cancer treatment (local or systematic) with either of the following:

     A. Pathologically confirmed gastric cancer diagnosis within 42 days prior to blood draw.

     B. High suspicious for cancer diagnosis by imaging tests or other routine clinical examinations, with confirmed pathological cancer diagnosis within 42 days after the blood draw.
  4. No peritoneal metastasis detected by laparoscopy with cytology.

Exclusion Criteria:

* Exclusion Criteria for All Participants:

  1. Insufficient qualified blood samples.
  2. During pregnancy or lactation.
  3. Recipient of organ transplant or prior non-autologous (allogeneic) bone marrow or stem cell transplant.
  4. Recipient of blood transfusion within 7 days prior to blood draw.
  5. Recipient of anti-tumor drugs to treat non-cancer diseases within 30 days prior to blood draw.
  6. With other known malignant tumors or multiple primary tumors.
* Exclusion Criteria for Control Arm Participants:

  1. Insufficient qualified blood samples.
  2. During pregnancy or lactation.
  3. Recipient of organ transplant or prior non-autologous (allogeneic) bone marrow or stem cell transplant.
  4. Recipient of blood transfusion within 7 days prior to blood draw.
  5. Recipient of anti-tumor drugs to treat non-cancer diseases within 30 days prior to blood draw.
  6. With other known malignant tumors or multiple primary tumors.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants of gastric cancer without any types of tumor treatment will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the cfDNA methylation-based model in detecting peritoneal metastasis of gastric cancer. | 30 months
Sensitivity and specificity of a cfDNA methylation-based model, in combination with other biomarkers, for detecting peritoneal metastasis of gastric cancer. | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Yihong Sun, Ph. D, Principal Investigator — Zhongshan Hospital, Fudan University, Shanghai, China; Xuefei Wang, Ph. D, Principal Investigator — Zhongshan Hospital, Fudan University, Shanghai, China
Locations (1):
- ZhongShan Hospital, Fudan university, Shanghai, China, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Thomassen I, van Gestel YR, van Ramshorst B, Luyer MD, Bosscha K, Nienhuijs SW, Lemmens VE, de Hingh IH. Peritoneal carcinomatosis of gastric origin: a population-based study on incidence, survival and risk factors. Int J Cancer. 2014 Feb 1;134(3):622-8. doi: 10.1002/ijc.28373. Epub 2013 Aug 5. PMID 23832847
- [Background] Allen CJ, Newhook TE, Vreeland TJ, Das P, Minsky BD, Blum M, Song S, Ajani J, Ikoma N, Mansfield PF, Roy-Chowdhuri S, Badgwell BD. Yield of peritoneal cytology in staging patients with gastric and gastroesophageal cancer. J Surg Oncol. 2019 Dec;120(8):1350-1357. doi: 10.1002/jso.25729. Epub 2019 Oct 14. PMID 31612494
- [Background] Chen M, Zhao H. Next-generation sequencing in liquid biopsy: cancer screening and early detection. Hum Genomics. 2019 Aug 1;13(1):34. doi: 10.1186/s40246-019-0220-8. PMID 31370908
- [Background] Kinoshita J, Fushida S, Harada S, Makino I, Nakamura K, Oyama K, Fujita H, Ninomiya I, Fujimura T, Kayahara M, Ohta T. Type IV collagen levels are elevated in the serum of patients with peritoneal dissemination of gastric cancer. Oncol Lett. 2010 Nov;1(6):989-994. doi: 10.3892/ol.2010.181. Epub 2010 Sep 23. PMID 22870099
- [Background] So JBY, Kapoor R, Zhu F, Koh C, Zhou L, Zou R, Tang YC, Goo PCK, Rha SY, Chung HC, Yoong J, Yap CT, Rao J, Chia CK, Tsao S, Shabbir A, Lee J, Lam KP, Hartman M, Yong WP, Too HP, Yeoh KG. Development and validation of a serum microRNA biomarker panel for detecting gastric cancer in a high-risk population. Gut. 2021 May;70(5):829-837. doi: 10.1136/gutjnl-2020-322065. Epub 2020 Oct 7. PMID 33028667
- [Background] Shimura T, Toden S, Kandimalla R, Toiyama Y, Okugawa Y, Kanda M, Baba H, Kodera Y, Kusunoki M, Goel A. Genomewide Expression Profiling Identifies a Novel miRNA-based Signature for the Detection of Peritoneal Metastasis in Patients With Gastric Cancer. Ann Surg. 2021 Nov 1;274(5):e425-e434. doi: 10.1097/SLA.0000000000003647. PMID 31663973
- [Background] Haber DA, Velculescu VE. Blood-based analyses of cancer: circulating tumor cells and circulating tumor DNA. Cancer Discov. 2014 Jun;4(6):650-61. doi: 10.1158/2159-8290.CD-13-1014. Epub 2014 May 6. PMID 24801577
- [Background] Pantel K, Alix-Panabieres C. Liquid biopsy and minimal residual disease - latest advances and implications for cure. Nat Rev Clin Oncol. 2019 Jul;16(7):409-424. doi: 10.1038/s41571-019-0187-3. PMID 30796368
- [Background] Qi C, Li P, Hu Y, et al. The ctDNA in peritoneal effusion of advanced gastric cancer for auxiliary diagnosis of peritoneal metastasis. Journal of Clinical Oncology. 2019/05/20 2019;37(15_suppl):e15516-e15516. doi:10.1200/JCO.2019.37.15_suppl.e15516
- [Background] Wu R, Li Q, Wu F, Shi C, Chen Q. Comprehensive Analysis of CDC27 Related to Peritoneal Metastasis by Whole Exome Sequencing in Gastric Cancer. Onco Targets Ther. 2020 Apr 21;13:3335-3346. doi: 10.2147/OTT.S244351. eCollection 2020. PMID 32368092
- [Background] Zhao D, Yue P, Wang T, Wang P, Song Q, Wang J, Jiao Y. Personalized analysis of minimal residual cancer cells in peritoneal lavage fluid predicts peritoneal dissemination of gastric cancer. J Hematol Oncol. 2021 Oct 12;14(1):164. doi: 10.1186/s13045-021-01175-2. PMID 34641926
- [Background] Klutstein M, Nejman D, Greenfield R, Cedar H. DNA Methylation in Cancer and Aging. Cancer Res. 2016 Jun 15;76(12):3446-50. doi: 10.1158/0008-5472.CAN-15-3278. Epub 2016 Jun 2. PMID 27256564
- [Background] Meng H, Cao Y, Qin J, Song X, Zhang Q, Shi Y, Cao L. DNA methylation, its mediators and genome integrity. Int J Biol Sci. 2015 Apr 8;11(5):604-17. doi: 10.7150/ijbs.11218. eCollection 2015. PMID 25892967
- [Background] Morgan AE, Davies TJ, Mc Auley MT. The role of DNA methylation in ageing and cancer. Proc Nutr Soc. 2018 Nov;77(4):412-422. doi: 10.1017/S0029665118000150. Epub 2018 Apr 30. PMID 29708096
- [Background] Widschwendter M, Jones A, Evans I, Reisel D, Dillner J, Sundstrom K, Steyerberg EW, Vergouwe Y, Wegwarth O, Rebitschek FG, Siebert U, Sroczynski G, de Beaufort ID, Bolt I, Cibula D, Zikan M, Bjorge L, Colombo N, Harbeck N, Dudbridge F, Tasse AM, Knoppers BM, Joly Y, Teschendorff AE, Pashayan N; FORECEE (4C) Consortium. Epigenome-based cancer risk prediction: rationale, opportunities and challenges. Nat Rev Clin Oncol. 2018 May;15(5):292-309. doi: 10.1038/nrclinonc.2018.30. Epub 2018 Feb 27. PMID 29485132
- [Background] Guo S, Diep D, Plongthongkum N, Fung HL, Zhang K, Zhang K. Identification of methylation haplotype blocks aids in deconvolution of heterogeneous tissue samples and tumor tissue-of-origin mapping from plasma DNA. Nat Genet. 2017 Apr;49(4):635-642. doi: 10.1038/ng.3805. Epub 2017 Mar 6. PMID 28263317
- [Background] Liu MC, Oxnard GR, Klein EA, Swanton C, Seiden MV; CCGA Consortium. Sensitive and specific multi-cancer detection and localization using methylation signatures in cell-free DNA. Ann Oncol. 2020 Jun;31(6):745-759. doi: 10.1016/j.annonc.2020.02.011. Epub 2020 Mar 30. PMID 33506766
- [Background] Harada H, Soeno T, Nishizawa N, Washio M, Sakuraya M, Ushiku H, Niihara M, Hosoda K, Kumamoto Y, Naitoh T, Sangai T, Hiki N, Yamashita K. Prospective study to validate the clinical utility of DNA diagnosis of peritoneal fluid cytology test in gastric cancer. Cancer Sci. 2021 Apr;112(4):1644-1654. doi: 10.1111/cas.14850. Epub 2021 Feb 27. PMID 33576114
- [Background] Hu XY, Ling ZN, Hong LL, Yu QM, Li P, Ling ZQ. Circulating methylated THBS1 DNAs as a novel marker for predicting peritoneal dissemination in gastric cancer. J Clin Lab Anal. 2021 Sep;35(9):e23936. doi: 10.1002/jcla.23936. Epub 2021 Aug 13. PMID 34390026
- [Background] Juzenas S, Venkatesh G, Hubenthal M, Hoeppner MP, Du ZG, Paulsen M, Rosenstiel P, Senger P, Hofmann-Apitius M, Keller A, Kupcinskas L, Franke A, Hemmrich-Stanisak G. A comprehensive, cell specific microRNA catalogue of human peripheral blood. Nucleic Acids Res. 2017 Sep 19;45(16):9290-9301. doi: 10.1093/nar/gkx706. PMID 28934507
- [Background] Rijken A, Lurvink RJ, Luyer MDP, Nieuwenhuijzen GAP, van Erning FN, van Sandick JW, de Hingh IHJT. The Burden of Peritoneal Metastases from Gastric Cancer: A Systematic Review on the Incidence, Risk Factors and Survival. J Clin Med. 2021 Oct 23;10(21):4882. doi: 10.3390/jcm10214882. PMID 34768402